CLINICAL TRIAL: NCT00512473
Title: Growth Hormone (GH) Signaling in Vivo in Human Muscle and Adipose Tissue: Impact of Insulin, Substrate Background and gh Receptor Blockade
Brief Title: Growth Hormone Signaling in Vivo in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 20050113
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2007-08-07 (Estimated); Status verified 2007-08

CONDITIONS: Intracellular Signaling Peptides and Proteins
Keywords: GH, GH receptor blockade, GH signaling, insulin resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Human Growth Hormone; pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Placebo Comparator): I.v. saline for 8 hours
  Interventions: Drug: Saline infusion
- GH (Experimental): Growth hormone (0.5 mg s.c. at t = 0 hours)
  Interventions: Drug: Human Growth Hormone
- Pegvisomant (Experimental): Pegvisomant injection 30 mg 36 hours prior to the study
  Interventions: Drug: Pegvisomant

INTERVENTIONS:
Drug: Saline infusion — 0.9 % NaCl
  Arms: A
Drug: Human Growth Hormone — 0.5 mg genotropin administered as a bolus at t = 0
  Arms: GH
Drug: Pegvisomant — 30 mg Somavert administered at t = - 36 hours
  Arms: Pegvisomant

SUMMARY:
Objective: GH induces insulin resistance in muscle and fat and in vitro data indicate that this may involve crosstalk between the signaling pathways of the two hormones.

Aim: To investigate GH and insulin signaling in vivo in human muscle and fat tissue in response to GH, GH receptor blockade and insulin stimulation..

DETAILED DESCRIPTION:
The molecular mechanisms by which GH promotes insulin antagonism are still unclear. Stimulation of lipolysis could be of importance since high plasma FFA levels have been shown to interfere with insulin receptor signaling via inhibition of insulin-stimulated insulin receptor substrate (IRS)-1 associated phosphatidylinositol (PI) 3-kinase activity in human skeletal muscle, resulting in a decreased GLUT4 translocation and glucose transport (6). A recent study, however, was unable to document a suppression in the insulin-stimulated activity of either IRS-1 associated PI 3-kinase or the serin/threonin kinase Akt after GH administration to healthy humans, despite induction of lipolysis and insulin resistance (7). Other studies have shown that acute GH exposure induces insulin resistance in skeletal muscle rapidly and before the subsequent rise in plasma FFA (1;7;8). These observations indicate that GH may cause insulin resistance via a non-FFA mediated mechanism.

The predominant GH signal transduction cascade comprises activation of the GHR dimer, phosphorylation of JAK2 and subsequently activation of Stat5. The intact JAK2/Stat5 pathway is necessary for normal statural growth (9). There is animal and in vitro evidence to suggest that insulin and GH share post-receptor signaling pathways (10). Convergence has been reported at the levels of Stat5 and SOCS3 as well as on protein kinases comprising the major IR signaling pathway; IRS 1/2, PI 3-kinase, Akt and ERK 1/2 (11-14).

Pegvisomant is a GH analog and a competitive reversible GH receptor antagonist, which blocks peripheral GH signal transduction (15). Pegvisomant has been shown to inhibit the necessary conformational change of the GHR dimer and thus constitutes an optimal negative control in GH signaling studies.

The aim of this work was to further study GH signal transduction pathways in vivo in muscle and adipose tissue from healthy subjects in response to acute and more prolonged GH exposure as well as during hyperinsulinemia. The design also included administration of pegvisomant in an attempt to correct for spontaneous GH secretion.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy
* Not taking medication

Exclusion Criteria:

* Insulin resistance

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2005-09; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
GH-receptor signaling | hours

SECONDARY OUTCOMES:
Insulin sensitivity | hours

CONTACTS AND LOCATIONS:
Overall Officials: Lars C Gormsen, MD, Principal Investigator — Aarhus University Hospital, Department M
Locations (1):
- Medical Research Laboratories, Aarhus, Denmark

REFERENCES:
- [Result] Gormsen LC, Nielsen C, Gjedsted J, Gjedde S, Vestergaard ET, Christiansen JS, Jorgensen JO, Moller N. Effects of free fatty acids, growth hormone and growth hormone receptor blockade on serum ghrelin levels in humans. Clin Endocrinol (Oxf). 2007 May;66(5):641-5. doi: 10.1111/j.1365-2265.2007.02786.x. PMID 17492951
- [Derived] Gormsen LC, Nielsen C, Jessen N, Jorgensen JO, Moller N. Time-course effects of physiological free fatty acid surges on insulin sensitivity in humans. Acta Physiol (Oxf). 2011 Mar;201(3):349-56. doi: 10.1111/j.1748-1716.2010.02181.x. Epub 2010 Oct 11. PMID 20731625
- [Derived] Nielsen C, Gormsen LC, Jessen N, Pedersen SB, Moller N, Lund S, Jorgensen JO. Growth hormone signaling in vivo in human muscle and adipose tissue: impact of insulin, substrate background, and growth hormone receptor blockade. J Clin Endocrinol Metab. 2008 Jul;93(7):2842-50. doi: 10.1210/jc.2007-2414. Epub 2008 May 6. PMID 18460563